CLINICAL TRIAL: NCT03055208
Title: Early Stereotactic Gamma Knife Radiosurgery to Residual Tumor After Surgery of Newly Diagnosed Glioblastoma
Acronym: Gamma-GBM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: suspended due to low accrual rates
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Frank A. Giordano, Interim Head, Department of Radiation Oncology, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gamma-GBM
Record Dates: First submitted 2017-02-09; First posted 2017-02-16 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Radiosurgery; Gamma Knife
MeSH Terms: conditions — Glioblastoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiosurgery (Experimental): Following intraoperative confirmation of glioblastoma (frozen section):
  Early (24-72h post surgery) stereotactic ablation (gamma knife radiosurgery) of residual tumor (defined in early postoperative T1-weighted MRI scanning with and without contrast), followed by standard-of-care therapy (chemo-radiotherapy with 60 Gy external beam radiation therapy (EBRT) and 75 mg/m2/d temozolomide, followed by adjuvant chemotherapy with 150-200 mg/m2/d/cycle temozolomide in a 5/28 days schedule).
  Interventions: Radiation: gamma knife radiosurgery (15 Gy to 50% isodose)

INTERVENTIONS:
Radiation: gamma knife radiosurgery (15 Gy to 50% isodose) — Radiosurgery with a gamma knife resembles the application of a precisely focused, high single dose of ionizing irradiation.

SUMMARY:
Gamma GBM is a single-arm phase II trial that prospectively measures the progression-free survival time after addition of an early gamma knife boost to areas of residual tumor to standard-of-care (surgery, chemo-radiotherapy, chemotherapy).

DETAILED DESCRIPTION:
Glioblastomas are highly malignant brain tumors that recur about 6 months after treatment. Most recurrences develop at the edge of the surgical margin and a common reason for an early recurrence of a glioblastoma is when tumors are not completely resected. This may be the case when intraoperative neuro-monitoring indicates that further resection would impair certain motor functions. Physicians can identify residual tumor in early (24-72h after surgery) postoperative MRI scans and could treat these regions. However, this treatment would not be a part of the recommended standard of care and thus, any further treatment of this areas will need a clinical trial.

The aim of this trial is to evaluate if the use of another modality to deplete these areas of residual tumor identified in early postoperative MRI scans will provide a relevant benefit in terms of progression-free survival (which means a prolongation of the time that patients do not experience a re-growth of the tumor). The modality is termed "radiosurgery", which is a non-invasive technique to delete cells without using a blade but a highly focused beam of gamma rays.

The machine that focusses these rays (like a magnifying glass that can focus light), is called 'gamma knife'. Gamma knife radiosurgery is a safe and effective treatment for a plethora of malignant and benign brain tumors and the technique is used since the 1950s and there has been a continuous improvement of precision and patient comfort up to now.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Karnofsky performance status score ≥ 60
* histology must be glioblastoma (frozen sections during surgery)
* radiographic proof of residual tumor
* Informed consent
* adequate birth control (e.g., oral contraceptives)

Exclusion Criteria:

* any previous cranial radiotherapy
* histology inconclusive or low(er)-grade astrocytoma
* contraindications for chemo- or radiotherapy
* bleeding or clotting disorders
* contraindications for MRI or CT scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2023-05-09 (Estimated)

PRIMARY OUTCOMES:
Median Progression-Free Survival Time (PFS) | 2 years
  PFS is defined as the time span of initial diagnosis (i.e., the day of surgery) until tumor progression is confirmed in follow-up MRI scans. All scans will be assessed using modified Response Assessment in Neuro-Oncology (RANO) criteria or until death by any cause.

SECONDARY OUTCOMES:
Median Overall Survival Time (OS) | 2 years
  OS is defined as the time span of initial diagnosis (i.e., the day of surgery) until death by any cause.
Radiation-related (acute / early delayed / late) neurotoxicity | 2 years
  Assessed by regular neurological examinations
Incidence of symptomatic radionecrosis | 2 years
  Assessed by serial MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Giordano, MD, Principal Investigator — University Medical Center Mannheim
Locations (1):
- Department of Radiotherapy University Hospital Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No